CLINICAL TRIAL: NCT05319054
Title: A Feasibility, Multicentre Randomised Control Trial Assessing the Treatment Options for Patient With Major Low Anterior Resection Syndrome to Establish a Pathway Of Low Anterior Resection Syndrome Relief After Surgery
Brief Title: Pathway of Low Anterior Resection Syndrome Relief After Surgery: a Feasibility Study
Acronym: POLARiS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cardiff and Vale University Health Board (Other Government)
Collaborators: University of Leeds (Other); Aneurin Bevan University Health Board (Other); University Hospital Southampton NHS Foundation Trust (Other); Bowel Research UK (Unknown); The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 8238; 307764 (Other: IRAS)
Record Dates: First submitted 2022-04-01; First posted 2022-04-08 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2022-11

CONDITIONS: Low Anterior Resection Syndrome
Keywords: Sacral Neuromodulation; Transanal Irrigation; Trials within cohorts; Colorectal cancer; Quality of Life
MeSH Terms: conditions — Low Anterior Resection Syndrome; Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Trials within Cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort (No Intervention): Patients who have undergone colonic resection for colorectal cancer in the last 10 years. Patient reported outcome measures collected at 3-monthly intervals.
- Optimised Conservative Management (Active Comparator): Cohort participants who are identified as having 'major LARS' at any point are treated with Optimised Conservative Managements, consisting of medication, dietary advice, lifestyle advice and physiotherapy.
  Interventions: Other: Optimised Conservative Management
- Trans-Anal Irrigation (Active Comparator): Cohort participants who are identified as having 'major LARS' at any point are treated with Trans-anal irrigation, in additional to receiving optimised conservative management. Transanal irrigation system will be decided upon with the participant and procured locally.
  Interventions: Device: Trans-Anal Irrigation; Other: Optimised Conservative Management
- Sacral NeuroModulation (Active Comparator): Cohort participants who are identified as having 'major LARS' at any point are treated with Sacral Neuromodulation system, in addition to receiving optimised conservative management. Medtronic Interstim system will be used.
  Interventions: Device: Sacral NeuroModulation; Other: Optimised Conservative Management

INTERVENTIONS:
Device: Sacral NeuroModulation — Sacral Neuromodulation group will include up-to 20 patients with major LARS. Medtronic Interstim system will be used, including 2 week trial device.
  Arms: Sacral NeuroModulation
Device: Trans-Anal Irrigation — Trans-Anal irrigation group will include up-to 20 patients with major LARS. Specific system will be agreed with the patient, depending on eligibility and preference.
  Arms: Trans-Anal Irrigation
Other: Optimised Conservative Management — Optimised conservative management will include up-to 30 patients with major LARS. They will be provided with a resource booklet which includes dietary and lifestyle advice as well as exercises that can be undertaken independently.
  Arms: Optimised Conservative Management; Sacral NeuroModulation; Trans-Anal Irrigation

SUMMARY:
Currently, no standard exists for the treatment and management of Low Anterior Resection Syndrome (LARS)- a common disorder that affects patients who have had part of their bowel removed due to colorectal cancer. Decisions about which treatment patients receive is at the discretion of local clinicians, leading to a variation in both clinical practice and the outcomes of these patients. As a result, there is a need for research to assess what treatments are most effective in treating or managing LARS to establish a consensus and develop a treatment pathway in the UK. This study aims to assess the feasibility of undertaking such a trial utilising a novel 'trial within cohorts (TWiCs)' study design, with a view to informing the design of a full-scale trial.

DETAILED DESCRIPTION:
Rectal cancer (cancer of the lower part of the bowel) is one of the most prevalent forms of cancer, and affects approximately 14,000 people each year in the UK. The treatment for the majority of these patients is surgical removal of the affected part of the bowel, following which the bowel is joined back together. Some patients may also require chemotherapy and radiotherapy. One consequence of the treatment of bowel cancer is a severe form of bowel dysfunction called major Low Anterior Resection Syndrome (LARS).

LARS is a constellation of symptoms including incontinence to stool, urgency and frequency of bowel movements and incomplete evacuation; it is diagnosed using the LARS scoring tool. Major LARS can have a huge impact on the persons quality of life resulting in social isolation. Currently there are no guidelines for the management of LARS. The aim of the POLARiS study is to investigate three different treatments for major LARS; optimised conservative management, a combination of diet, medication, bowel retraining and pelvic floor exercises; transanal irrigation, washing out the back passage of stool with warmed water; and sacral nerve stimulation where an electrical impulse delivered to the sacral nerve to help with bowel function. This feasibility study aims to test the study design ahead of a larger fully powered randomised control trial. The study will firstly recruit any consenting adult who has had surgery for rectal cancer (called an anterior resection) and who does not have a stoma, into a cohort and then follow up those patients every 3 months with bowel function and quality of life assessments. Any patient found to have major LARS (LARS score over 30) will be invited into the randomised control trial where the above three treatments will be tested.

ELIGIBILITY:
Inclusion Criteria:

* For cohort:

  * Diagnosis of rectal or sigmoid cancer
  * Low or high anterior resection (colorectal resection with anastomosis to the rectum)
  * Functioning anastomosis
  * Aged 18 years and older
  * Primary surgery/reversal of ileostomy less than 10 years before recruitment
  * Reversal of ileostomy at least 12 weeks prior to recruitment with at least a further 12 weeks of standard care to manage symptoms following reversal
  * Willing and able to provide valid informed consent
* For randomisation:

  * Recruited to cohort study
  * Willing and able to provide valid informed consent for randomisation
  * Major LARS symptoms (Defined as score of 30+ on LARS scoring tool)
  * Previous unsuccessful conservative treatment determined by treating clinician and patient

Exclusion Criteria:

* For cohort

  - Inability to understand and complete study questionnaires independently. (Due to cognitive or intellectual impairment, Due to insufficient English language skills)
* For randomised control trial

  * Pregnancy
  * No previous conservative treatment plan for the management of LARS
  * Does not meet any treatment-specific criteria
* For TAI randomisation:

  * Unable to perform TAI
  * History of anastomotic leak with evidence of ongoing leak/sinus
  * Previous use of TAI for LARS
  * Site unable to offer TAI as a treatment
  * Any other contraindications advised by the care team, product manufacturer or distributor
* For SNM randomisation:

  * <12months since primary cancer surgery
  * Palliative disease
  * Site unable to offer SNM as a treatment
  * Previous SNM
  * Specific contraindications to implantation
  * Any other contraindications advised by the care team, product manufacturer or distributor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate of to cohort arm of study | 9 months
  The total number of participants enrolled into the study over the recruitment period.
Assess characteristics of patients recruited to the cohort | 9 months
  We will record basic demographics, medical history and prevalence of relative symptoms of participants enrolled in the cohort study to describe the characteristics of no- minor- and major- LARS patients
Prevalence of 'major LARS' in the patient cohort | 12 months
  The number of participants in the cohort that meet the criteria for 'major low anterior resection syndrome (LARS)', as measured by the LARS scoring tool. LARS scoring tool produces a score from 0 - 42, which represents the severity of symptoms, where 0 is least severe and 42 is most severe. Score =>30 is considered 'major LARS'. LARS score will be measured at 5 times at 3-monthly intervals over 12 months.
Onset of 'major LARS' symptoms in relation to surgery | Time from surgery to onset of major LARS, up to 10 years.
  The time (in months) from resection surgery to onset of 'major LARS' symptoms, as reported by the LARS scoring tool.
Onset of 'major LARS' symptoms in relation to radiotherapy treatment | Time from ending radiotherapy treatment to onset of major LARS, up to 10 years.
  The time (in months) from completing radiotherapy treatment to onset of 'major LARS' symptoms, as reported by the LARS scoring tool.
Recruitment rate to randomised trial part of the study | 9 months
  The total number of cohort participants that are enrolled into the randomised trial part of the study, over the recruitment period.
Proportion of randomised participants that are allocated to each trial arm | 9 months
  The proportion of randomised participants that meet the criteria for, and are allocated to, each of the three trial arms (transanal irrigation; sacral neuromodulation; optimised conservative management).
Describe variation in clinical practice across UK sites | Up to 10 years prior to recruitment
  Where possible, we will record patient's previous treatments and interactions with health services in relation to their bowel dysfunction symptoms. This will be used to describe the variation in UK clinical practice in terms of diagnosis, management and treatment pathways.
Compliance of participants to the study programme | 12 months
  The proportion of participants that complete and return follow-up questionnaires (four questionnaires at 3-month intervals).
Adherence of participants to the treatment programme | 12 months
  The proportion of patients that continue to receive the treatment assigned to them at the end of the follow-up period.

SECONDARY OUTCOMES:
Change in LARS score | 12 months.
  LARS score will be measured at 5 time points (at 3-monthly intervals from baseline to 12 months) to assess severity of bowel dysfunction. Self-reported by participants using the LARS scoring tool (min 0, max 42) where higher score denotes greater severity of symptoms.
Change in EuroQuol 5-Dimension Health-related Quality of Life instrument (5-level) (EQ-5D-5L) | 12 months
  Patient-reported quality of life will be measured using the EuroQuol 5-Dimension Health-related Quality of Life instrument (5-level) (EQ-5D-5L) at 5 time-points (3-monthly intervals from baseline to 12 months). Quality of life total score will be calculated (min 5; max 25), where reduction in total score represents improvement in quality of life.
Change in European Organisation for Research and Treatment of Cancer Colorectal Quality of Life Questionnaire | 12 months
  Quality of life will be self-reported by participants using the European Organisation for Research and Treatment of Cancer Colorectal Quality of Life Questionnaire (EORTC QLQ-CR29) at 5 time-points (3-monthly intervals, from baseline to 12 months). Quality of life total score will be calculated (min 26; max 104) where reduction in total score represents improvement in quality of life.
Change in European Organisation for Research and Treatment of Cancer Cancer Quality of Life Questionnaire | 12 months
  Quality of life will be self-reported by participants using the European Organisation for Research and Treatment of Cancer Cancer Quality of Life Questionnaire (EORTC QLQ-C30). This will be recorded at 5 time-points (3-monthly intervals, from baseline to 12 months). Total score will be calculated (min 30; max 128), where reduction in total score represents improvement in quality of life.
Change in medical outcome profile score | 12 months
  Measure Yourself Medical Outcome Profile (MYMOP) 2 will be used to record patient-reported medical outcome profile at 5 time-points (3-montly intervals from baseline to 12 months). Change in patient-reported severity (min 0; max 5) will be measured, where change ≥ 1.0 is considered clinically significant.
Patient-reported adverse events | 12 months
  We will record any adverse events reported by randomised patients in relation to each of the treatments they receive, which impairs their adherence to the study protocol, treatment programme or safety.
LARS treatment history | 12 months
  Treatments offered to manage individual patient's LARS symptoms will be recorded, along with duration of treatment and reasons for stopping. This will be used to support the description of standard care variation and patient characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Cornish, Principal Investigator — Cardiff and Vale University Health Board
Locations (4):
- United Kingdom (4):
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - Leeds Teaching Hospital NHS Trust, Leeds, Yorkshire
  - Julie Cornish, Cardiff
  - Royal Gwent Hospital, Newport

IPD SHARING:
Plan to Share IPD: No